CLINICAL TRIAL: NCT02005731
Title: A Prospective Multicenter Pilot Study to Assess the Safety and Efficacy of Low Intensity Extracorporeal Shockwave Therapy (LI-ESWT) by 'Renova' in Patients With Erectile Dysfunction
Brief Title: Low Intensity Extracorporeal Shockwave Therapy for Patients With Erectile Dysfunction
Acronym: LISW
Status: Completed | Type: Observational
Sponsor: Initia (Industry)
Responsible Party: Sponsor
Other Study IDs: LSWT-004-EU
Record Dates: First submitted 2013-12-04; First posted 2013-12-09 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Vasculogenic Erectile Dysfunction
Keywords: Low Intensity Shockwave; Extracorporeal shockwave therapy; Erectile dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Shockwaves: Low intensity linear focused shockwave device ('Renova')
  Interventions: Device: Low intensity linear focused shockwave device ('Renova')

INTERVENTIONS:
Device: Low intensity linear focused shockwave device ('Renova')

SUMMARY:
This is a prospective, pilot study for assessing the safety and efficacy of the treatments performed with Renova (LI-ESWT) on symptomatic ED patients.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Vasculogenic ED for at least 6 months
* International Index of Erectile Function 6 (IIEF-EF) between 11 to 25
* Positive response to PDE5-I (able to penetrate on demand, Responders)
* Negative response to PDE5-I (unable to penetrate on demand even with maximum PDE5-I dosage,Non-responders)
* Stable heterosexual relationship for more than 3 months

Exclusion Criteria:

* Psychogenic ED
* Neurological pathology
* Hormonal pathology
* Past radical prostatectomy
* Recovering from cancer during last 5 years
* Any unstable medical, psychiatric, spinal cord injury and penile anatomical - abnormalities
* Clinically significant chronic hematological disease
* Anti-androgens, oral or injectable androgens
* Radiotherapy in pelvic region

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sexual Medicine clinic
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the IIEF-EF (International Index of Erectile Function- Erectile Function Domain) score at 1, 3 and 6 months post treatment | 1, 3 and 6 months post treatment

SECONDARY OUTCOMES:
Change from baseline in the SEP (Sexual Encounter Profile) Questions 2 and 3 at 1, 3 and 6 months post treatment | 1, 3 and 6 months post treatment
Responses to the GAQ (Global Assessment questions) Questions 1 and 2 at 1, 3 and 6 months post treatment | 1, 3 and 6 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Cobi Reisman, MD, PhD, Principal Investigator — Men's Health Clinic, Amstelland Hospital, Amsterdam, The Netherlands
Locations (4):
- Urologickaambulance, Brno, Czechia
- Amber Clinic, Klaipėda, Lithuania
- Men's Health Clinic, Amstelland Hospital, Amsterdam, Netherlands
- Urology and Andrology Center, Red Crescent Hospital (RCH), Ramallah, Palestinian Territories

REFERENCES:
- [Background] Vardi Y, Appel B, Jacob G, Massarwi O, Gruenwald I. Can low-intensity extracorporeal shockwave therapy improve erectile function? A 6-month follow-up pilot study in patients with organic erectile dysfunction. Eur Urol. 2010 Aug;58(2):243-8. doi: 10.1016/j.eururo.2010.04.004. Epub 2010 May 6. PMID 20451317
- [Background] Goyal NK, Garg M, Goel A. Re: Does low intensity extracorporeal shock wave therapy have a physiological effect on erectile function? Short-term results of a randomized, double-blind, sham controlled study: Y. Vardi, B. Appel, A. Kilchevsky and I. Gruenwald. J Urol 2012; 187: 1769-1775. J Urol. 2012 Nov;188(5):2018-9. doi: 10.1016/j.juro.2012.07.052. Epub 2012 Sep 20. No abstract available. PMID 22999553
- [Background] Rosen RC, Cappelleri JC, Gendrano N 3rd. The International Index of Erectile Function (IIEF): a state-of-the-science review. Int J Impot Res. 2002 Aug;14(4):226-44. doi: 10.1038/sj.ijir.3900857. PMID 12152111
- [Background] Rosen RC, Allen KR, Ni X, Araujo AB. Minimal clinically important differences in the erectile function domain of the International Index of Erectile Function scale. Eur Urol. 2011 Nov;60(5):1010-6. doi: 10.1016/j.eururo.2011.07.053. Epub 2011 Jul 30. PMID 21855209